CLINICAL TRIAL: NCT04998136
Title: Efficacy and Safety of Semaglutide 2.4 mg Once-weekly in Asians With Obesity Diagnosed as BMI ≥ 25 kg/m2 According to Local Guidelines
Brief Title: Research Study Investigating How Well Semaglutide Works in People From Thailand and South Korea Living With Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4707; U1111-1265-5285 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide 2.4 mg (Experimental)
  Interventions: Drug: Semaglutide 2.4 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (semaglutide 2.4 mg)

INTERVENTIONS:
Drug: Semaglutide 2.4 mg — Administered subcutaneously (s.c., under the skin) as well as reduced-calorie diet and increased physical activity for 44 weeks. Doses gradually increased to 2.4 mg
  Arms: Semaglutide 2.4 mg
Drug: Placebo (semaglutide 2.4 mg) — Administered s.c. as well as reduced-calorie diet and increased physical activity for 44 weeks
  Arms: Placebo

SUMMARY:
This study looks at how well semaglutide helps people lose weight. This study will look at the change in the participants' body weight from the start to the end of the study. The study compares the weight loss in people who get semaglutide to the weight loss in people who get placebo. Placebo is a "dummy" medicine that looks like the study medicine, but has no effect on the body.

Participants will either get semaglutide or "dummy" medicine - which treatment participants get is decided by chance. Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm.

Participants will also have talks with study staff about healthy food choices, how to be more physically active and what participants can do to lose weight.

The study will last for about a year (50 weeks). Participants will have 10 clinic visits and 8 phone calls. At 6 of the clinic visits participants will have blood samples taken.

Participants cannot take part if participants have or have had diabetes. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years at the time of signing informed consent.
* BMI at least 25.0 kg/m^2 at screening.
* Both parents of Asian descent.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* HbA1c at least 48 mmol/mol (6.5%) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes mellitus.
* A self-reported change in body weight above 5 kg (11 lbs) within 90 days before screening irrespective of medical records.
* Any participant where a substantial weight loss, in the investigator's opinion, might jeopardise the participant's safety.
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) below 15 mL/min/1.73 m^2 at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (16):
- South Korea (7):
  - Konyang University Hospital, Daejeon
  - Dongguk University Ilsan Hospital_Gyeonggi-do, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Thailand (9):
  - King Chulalongkorn Memorial Hospital_Bangkok, Bangkok
  - King Chulalongkorn Memorial Hospital_Endocrinology, Bangkok
  - King Chulalongkorn Memorial Hospital_Obstetrics&Gynecology, Bangkok
  - Obstetrics&Gynecology King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital_Nutrition and Biochemical, Bangkok
  - Siriraj Hospital_Bangkok_1, Bangkok
  - Siriraj Hospital_Dept Cardio, Bangkok
  - Siriraj Institute of Clinical Research, Bangkok
  - Maharaj Nakorn Chiang Mai_Hematology and Oncology, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Lim S, Buranapin S, Bao X, Quiroga M, Park KH, Kang JH, Rinnov AR, Suwanagool A. Once-weekly semaglutide 2.4 mg in an Asian population with obesity, defined as BMI >/=25 kg/m2, in South Korea and Thailand (STEP 11): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2025 Oct;13(10):838-847. doi: 10.1016/S2213-8587(25)00164-0. Epub 2025 Aug 15. PMID 40825340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 13 sites in Republic of Korea and Thailand.
Pre-assignment Details: The trial included an initial 16 weeks of dose escalation period and a 28 weeks of maintenance period. 150 eligible participants were randomized in a 2:1 manner to receive either Semaglutide or placebo once weekly as an adjunct to a reduced-calorie diet and increased physical activity.
Groups:
- Semaglutide: Participants received 2.4 milligram (mg) semaglutide subcutaneous injection once weekly using PDS290 pen injector for 44 weeks. Participants initially received (0.25 mg) semaglutide once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (2.4 mg) was reached: 0.25 mg (week 1 - week 4), 0.5 mg (week 5 - week 8), 1.0 mg (week 9 - week 12), 1.7 mg (week 13 - week 16), 2.4 mg (week 17 - week 44). The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
- Placebo: Participants received placebo matched to semaglutide once weekly by subcutaneous injection for 44 weeks. Participants initially received 0.25 mg placebo matched to semaglutide once weekly and the dose was then escalated once in 4 weeks until maintenance dose was reached: 0.25 mg (week 1- week 4), 0.5 mg (week 5 - week 8), 1.0 mg (week 9 - week 12), 1.7 mg (week 13 - week 16), 2.4 mg (week 17 - week 44). The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
Period: Overall Study
Arm/Group | Semaglutide | Placebo
Started | 101 | 49
Full Analysis Set | 101 | 49
Safety Analysis Set | 101 | 49
Completed | 101 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Semaglutide: Participants received 2.4 mg semaglutide subcutaneous injection once weekly using PDS290 pen injector for 44 weeks. Participants initially received (0.25 mg) semaglutide once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (2.4 mg) was reached: 0.25 mg (week 1 - week 4), 0.5 mg (week 5 - week 8), 1.0 mg (week 9 - week 12), 1.7 mg (week 13 - week 16), 2.4 mg (week 17 - week 44). The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Placebo | Total
Number analyzed (Participants) | 101 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (10) | 37 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 33 | 111
  Male | 23 | 16 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 49 | 150
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 101 | 49 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%) : In-trial Observation Period
Description: Change in percentage (%) of body weight from baseline (week 0) to end of treatment (week 44) is presented in this outcome measure and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial observation period: The time period where the participants were assessed in the study. The in-trial observation period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: FAS included all randomized participants. Here, Overall number of participants analysed (N) = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Percentage of body weight | -16.4 (7.3) | -2.6 (5.8)
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Treatment policy Estimand. The primary endpoint was analysed using an analysis of covariance (ANCOVA) model with randomized treatment as factor and baseline body weight as covariate. Analysed data is from in-trial observation period; Test type: Superiority; p < 0.0001, ANCOVA; Treatment difference = -12.99, 95% CI 2-sided [-15.28 to -10.70]

2. Primary Outcome: Change in Body Weight (%) : On-treatment Observation Period
Description: Change in percentage (%) of body weight from baseline (week 0) to end of treatment (week 44) is presented in this endpoint. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: The time period where participants were treated with trial product. It started from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) including 2 weeks of follow up. It excludes off treatment period which is defined as at least 2 consecutive missed doses.
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 96 | 47
Percentage of body weight | -16.4 (7.4) | -2.7 (5.8)
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Hypothetical Estimand. The primary endpoint was analysed using mixed model for repeated measurements (MMRM). All responses prior to first discontinuation of treatment (or dose reduction, or initiation of other anti-obesity medication or bariatric surgery) were included in MMRM with randomized treatment as factor and baseline body weight as covariate. Analysed data is from on-treatment observation period; Test type: Superiority; p < 0.0001, MMRM; Treatment Difference = -13.40, 95% CI 2-sided [-15.70 to -11.11]

3. Primary Outcome: Number of Participants Achieved More Than or Equal to (≥) 5 Percent (%) Body Weight Reduction (Yes/no) : In-trial Observation Period
Description: Number of participants who achieved body weight reduction more than or equal to 5 percent is presented at week 44 in this outcome measure and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial observation period: The time period where the participants were assessed in the study. The in-trial observation period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: At week 44
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Participants
  Yes | 96 | 12
  No | 4 | 36
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Treatment policy estimand. The primary endpoint was analysed using a binary logistic regression model with randomized treatment as factor and baseline body weight as covariate. Analysed data is from in-trial period; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 88.87, 95% CI 2-sided [21.96 to 359.61]

4. Primary Outcome: Number of Participants Achieved More Than or Equal to (≥) 5 Percent (%) Body Weight Reduction (Yes/no) : On-treatment Observation Period
Description: Number of participants who achieved body weight reduction more than or equal to 5 percent is presented at week 44 in this endpoint. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: the time period where partici-pants were treated with trial product. It started from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) including 2 weeks of follow up. It excludes off treatment period which is defined as at least 2 consecutive missed doses.
Time Frame: At week 44
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 96 | 47
Participants
  Yes | 92 | 12
  No | 4 | 35
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Hypothetical estimand. MMRM was used with randomized treatment as factor and baseline body weight as covariate. The MMRM was performed on body weight (kg) and individual missing week 44 responses were predicted from the MMRM, each participant was then classified for body weight loss >= 5% and analysed using a binary logistic regression model with randomized treatment as factor and baseline body weight as covariate. Analysed data is from on-treatment observation period; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 253.47, 95% CI 2-sided [38.41 to 1672.57]

5. Secondary Outcome: Number of Participants Achieved ≥ 10% Body Weight Reduction (Yes/no)
Description: Number of participants who achieved body weight reduction more than or equal to 10 percent is presented at week 44 and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: At week 44
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Participants
  Yes | 78 | 5
  No | 22 | 43

6. Secondary Outcome: Number of Participants Achieved ≥15% Body Weight Reduction (Yes/no)
Description: Number of participants who achieved body weight reduction more than or equal to 15 percent is presented at week 44 and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: At week 44
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Participants
  Yes | 53 | 2
  No | 47 | 46

7. Secondary Outcome: Number of Participants Achieved ≥20% Body Weight Reduction (Yes/no)
Description: Number of participants who achieved body weight reduction more than or equal to 20 percent is presented at week 44 and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: At week 44
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Participants
  Yes | 30 | 0
  No | 70 | 48

8. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to the end of treatment (week 44) is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Centimeter (cm) | -12.0 (7.5) | -3.0 (5.4)

9. Secondary Outcome: Change in Body Weight (kg)
Description: Change in body weight in kilogram (kg) is presented from baseline (week 0) to the end of treatment (week 44) and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Kg | -13.0 (5.5) | -2.0 (5.1)

10. Secondary Outcome: Change in Body Mass Index
Description: Change in body mass index from baseline (week 0) to end of treatment (week 44) is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Kilogram per square meter (kg/m^2) | -4.9 (2.1) | -0.8 (1.9)

11. Secondary Outcome: Change in Systolic Blood Pressure (mmHg)
Description: Change in systolic blood pressure from baseline (week 0) to end of treatment (week 44) is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Millimeter of mercury (mmHg) | -11 (14) | -1 (13)

12. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to end of the treatment (week 44) is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: MmHg
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
MmHg | -4 (11) | 0 (12)

13. Secondary Outcome: Change in Total Cholesterol (mg/dL) - Ratio to Baseline
Description: Change in total cholesterol in milligram per deciliter (mg/dL) from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Ratio of total cholesterol | 0.91 (15.7) | 1.03 (12.3)

14. Secondary Outcome: Change in Total Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in total cholesterol in millimoles per liter (mmol/L) from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Ratio of total cholesterol | 0.91 (15.7) | 1.03 (12.3)

15. Secondary Outcome: Change in High-density Lipoprotein (HDL) Cholesterol (mg/dL) - Ratio to Baseline
Description: Change in HDL cholesterol in mg/dL from (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 99 | 48
Ratio of HDL cholesterol | 1.00 (15.3) | 1.04 (13.7)

16. Secondary Outcome: Change in High-density Lipoprotein (HDL) Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in HDL cholesterol in mmol/L from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 99 | 48
Ratio of HDL cholesterol | 1.00 (15.3) | 1.04 (13.7)

17. Secondary Outcome: Change in Low-density Lipoprotein (LDL) Cholesterol (mg/dL) - Ratio to Baseline
Description: Change in LDL cholesterol in mg/dL from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 99 | 48
Ratio of LDL cholesterol | 0.93 (25.6) | 1.04 (21.6)

18. Secondary Outcome: Change in Low-density Lipoprotein (LDL) Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in LDL cholesterol in mmol/L from baseline (week 0) to end of treatment (week 44) as ratio to baseline presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 99 | 48
Ratio of LDL cholesterol | 0.93 (25.6) | 1.04 (21.6)

19. Secondary Outcome: Change in Triglycerides (mg/dL) - Ratio to Baseline
Description: Change in triglycerides in mg/dL from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Ratio of triglycerides | 0.72 (40.9) | 0.96 (42.1)

20. Secondary Outcome: Change in Triglycerides (mmol/L) - Ratio to Baseline
Description: Change in triglycerides in mmol/L from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Ratio of triglycerides | 0.72 (40.9) | 0.96 (42.1)

21. Secondary Outcome: Change in High-sensitivity C-reactive Protein (hsCRP) (mg/L) - Ratio to Baseline
Description: Change in hsCRP in milligram per liter (mg/L) from baseline (week 0) to end of treatment (week 44) as ratio to baseline is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 48
Ratio of hsCRP | 0.54 (170.0) | 0.89 (73.7)

22. Secondary Outcome: Change in HbA1c (%)
Description: Change in glycosylated haemoglobin (HbA1c) in percentage from baseline (week 0) to end of treatment (week 44) is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 47
Percentage of HbA1c | -0.4 (0.3) | 0.0 (0.2)

23. Secondary Outcome: Change in HbA1c (mmol/Mol)
Description: Change in glycosylated heamoglobin (HbA1c) in millimoles per mole (mmol/mol) from baseline (week 0) to end of treatment (week 44) is presented and it was evaluated based on the data from in-trial observation period. For end of treatment visit, data collected up to week 49 during the in-trial observation period is included in this Outcome Measure. In-trial period: The time period where the participants were assessed in the study. The in-trial period begins on the date of randomization (week 0) and ends at the end of study visit (week 49).
Time Frame: Baseline (week 0), end of treatment (week 44)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mmol/mol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 100 | 47
Mmol/mol | -4.5 (3.2) | -0.1 (2.3)

ADVERSE EVENTS:
Time Frame: From (week 0) to (week 49).
Description: All presented AEs are TEAEs (treatment emergent adverse events).
  Adverse events will be defined as "treatment-emergent" (TEAE), if the onset of the event occurs in the on-treatment period.
  Safety analysis set (SAS): All participants who were exposed to at least one dose of randomised IMP. Participants were included in the analyses according to the intervention they actually received.
Arm/Group | Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/49
Serious Adverse Events (participants affected / at risk) | 13/101 | 4/49
Other Adverse Events (participants affected / at risk) | 80/101 | 34/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=101) | Placebo (N=49)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Chikungunya virus infection (Infections and infestations) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=101) | Placebo (N=49)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
COVID-19 (Infections and infestations) | 15 (17) | 16 (16)
Constipation (Gastrointestinal disorders) | 22 (24) | 8 (10)
Decreased appetite (Metabolism and nutrition disorders) | 13 (14) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 28 (43) | 3 (3)
Dizziness (Nervous system disorders) | 11 (13) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 12 (18) | 5 (5)
Gastroenteritis (Infections and infestations) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 13 (20) | 3 (7)
Nasopharyngitis (Infections and infestations) | 12 (16) | 12 (17)
Nausea (Gastrointestinal disorders) | 38 (57) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 7 (10)
Vomiting (Gastrointestinal disorders) | 11 (13) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT04998136/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT04998136/SAP_001.pdf